CLINICAL TRIAL: NCT00517114
Title: Prospective Double-blinded Randomized Controlled Trial of 12-weeks High Dose Rabeprazole (Pariet) in the Treatment of Reflux Laryngitis in Chinese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW04-204 T/526; HARECCTR0500033
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Gastroesophageal Reflux; Laryngitis
Keywords: Reflux laryngitis
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngitis | interventions — Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole 20mg twice daily

SUMMARY:
The purpose of this study is to evaluate the efficacy of rabeprazole (pariet) versus placebo in treating reflux laryngitis in Chinese patients. Patients who attend the voice clinic of Department of ENT, Queen Mary hospital with suspected reflux laryngitis will be recruited. A questionnaire will be administered by the research assistant of the Department of Medicine and ENT, Queen Mary hospital. A 12-week course of PPI versus placebo trial will be commenced and patients' symptoms and signs will be documented at 6-week and 12-week time. The study will finish after a 12-week course of rabeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with age between 18-80 years old
* Patients with newly presented laryngitis.

Exclusion Criteria:

* They were under 18 or over 80 years of age
* Has significant concomitant medical disease
* Pregnancy or lactating women
* Chronic cough attributable to known chronic pulmonary or tracheobronchial disease
* Previous glottal surgery, radiotherapy or malignancy
* Acid suppressive therapy within 4 wk prior to recruitment
* Pharyngo-laryngeal infection in the previous 3 months
* Tracheal intubation in previous 12 months
* Immunosuppression and use of inhaled corticosteroid

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-01; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Symptoms assessment, quality of life. | 12 weeks

SECONDARY OUTCOMES:
Compliance | 4 weeks
Adverse effects | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul KY Lam, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China